CLINICAL TRIAL: NCT06223321
Title: The Role of Multislice Computed Tomography in Congenital Heart Diseases in Paediatric Age Group.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Collaborators: Magdi Yacoub Heart Foundation (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdelghany Elsherif, ASSISTANT LECTURE AT DIAGNOSTIC AND INTERVENTIONAL RADIOLOGY DEPARTMENT, Sohag University
Other Study IDs: Soh-Med-23-12-02MD
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Congenital Heart Diseases
Keywords: Computed Tomography - congenital heart diseases
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Computed Tomography in congenital heart diseases — ● CT examination will be done by
  * 160 MDCT Toshiba Machine or 128 MDCT GE machine or 160 MDCT Philips Machine:
  * We used the following parameters during cardiac CT scanning:
    * Pitch of 1.3, helical thickness of 0.5 mm and coverage of 32 cm.
    * The radiation dose set to 80-100 kvp.
    * Tube current from 10 to 40 mA/kg.
    * The gantry rotation speed at 0.35-.4 sec.
    * ECG gated Retrospective With MA modulation.
    * Wide FOV.
  * A scout will be taken and dual-phase injection conducted using non ionized contrast material. The total contrast volume is 1.5-3 ml/kg.
  * Scanning begins when contrast filled the LV by bolus tracking.
  * All images were transferred to workstation multiplanar reformation (MPR), maximum (MIP) and minimum (MinIP) intensity projections and volume rendering images will be performed for reporting.

SUMMARY:
This study aims to evaluate the added value of cardiac multislice Computed Tomography in assessment of CHD in pediatrics as a non-invasive presurgical planning method

DETAILED DESCRIPTION:
All patients will be subjected to the followings:

* All children gave an informed consent prior performing the research.
* Every child was submitted to full history taking.
* Clinical assessment of the patients will be performed in the form of: measuring of vital signs and anthropometric measurements.
* Renal function tests(ѕerum creatinine and blood urea).
* Patients will be prepared for CT as following:

  * Calculation of amount of CM and sedations.
  * The patient will be fasting for 4 hours.
  * The peripheral venous line will placed usually in a right upper limb vein, exercise if cosurgical .
  * The patients will be put in a supine position and at the middle of CT gantry.
  * ECG leads will be put on the chest of the patient. Infants below 6 months will be laid with arms at their side or above their head for image acquisition, positioning the arms above their head is advised, while patients above 6 months of age were positioned with their arms above their head when possible.
* CT examination will be done by

  * 160 MDCT Toshiba Machine or 128 MDCT GE machine or 160 MDCT Philips Machine:
  * We used the following parameters during cardiac CT scanning:

    * Pitch of 1.3, helical thickness of 0.5 mm and coverage of 32 cm.
    * The radiation dose set to 80-100 kvp.
    * Tube current from 10 to 40 mA/kg.
    * The gantry rotation speed at 0.35-.4 sec.
    * ECG gated Retrospective With MA modulation.
    * Wide FOV.
  * A scout will be taken and dual-phase injection conducted using non ionized contrast material. The total contrast volume is 1.5-3 ml/kg.
  * Scanning begins when contrast filled the LV by bolus tracking.
  * All images were transferred to workstation multiplanar reformation (MPR), maximum (MIP) and minimum (MinIP) intensity projections and volume rendering images will be performed for reporting.
  * Reporting in sequential approach

    * Cardiac sidedness
    * Cardiac position
    * Three segments , atrial chambers , ventricular chambers and the great arteries (aorta and pulmonary arteries)
    * Cardiac connections (veno-atrial ,atrio-ventricular and ventriculo-arterial )
    * Associated malformation (intra cardiac communications , valvular pathologies)
    * Aortic arch and its branching pattern
    * Pulmonary arteries
    * Pulmonary veins (number and drainage pattern )
    * SVC,IVC (their course and draining pattern )
    * Systematic veins azygos , hemiazygos and brachiocephalic vein
    * Coronary arteries
    * Position of abdominal organs( liver spleen, stomach & pancrease )
    * Secondary changes in cardiac chambers and lung parenchyma
    * Bony anomalies
  * Results: Results will be tabulated and assessed statistically and compared to other published results.
  * Ethical consideration and Study approval: The study protocol will be approved by the ethics committee of Faculty of Medicine, Sohag University.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suspected to have congenital heart disease based on clinical findings.
2. Patients known to have congenital heart diseased based on echocardiography (ECHO) with ECHO findings are not sufficient and referred to perform CT for further assessment

Exclusion Criteria:

* Post-operative Patients of congenital heart disease.
* Patients who are known to have hyper susceptibility to iodinated Contrast media reaction, impaired renal functions, respiratory failure, fever and severe asthma and patients with arrhythmia.

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: * All children gave an informed consent prior performing the research.
  * Every child was submitted to full history taking.
  * Clinical assessment of the patients will be performed in the form of: measuring of vital signs and anthropometric measurements.
  * Renal function tests(ѕerum creatinine and blood urea).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Multislice Computed Tomography in congenital heart diseases in Paediatric age group | within one week after Computed Tomography done
  added value of cardiac multislice Computed Tomography in assessment of CHD in pediatrics as a non-invasive presurgical planning method (detection of other lesion not seen by other imaging modalities )

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AA Elsherif, ASSISST. LEC, Principal Investigator — Sohag University Hospitals
Locations (1):
- Sohag university hospitals- faculity of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided